CLINICAL TRIAL: NCT05060133
Title: Changes of the Upper Airway Volume After Orthognathic Surgery - is This a Treatment Option of Severe Obstructive Sleep Apnea?
Brief Title: Changes of the Upper Airway Volume After Orthognathic Surgery
Status: Completed | Type: Observational
Sponsor: Lund University Hospital (Other)
Responsible Party: Principal Investigator, Martin Bengtsson, Consultant Oral and Maxillofacial Surgeon, Lund University Hospital
Other Study IDs: OFRS939554
Record Dates: First submitted 2021-09-13; First posted 2021-09-29 (Actual); Last update posted 2023-01-30 (Actual); Status verified 2023-01

CONDITIONS: OSA; Malocclusion; Dentofacial Deformities
MeSH Terms: conditions — Malocclusion; Dentofacial Deformities | interventions — Orthognathic Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Orthognathic Surgery — Surgical corrections of dentofacial deformities and malocclusions.

SUMMARY:
The aim of the present project is to analyze the impact from orthognathic surgery on the upper airway respiratory volume.

The primary objective is comparison of differences in the in the airway changes due to maxillary movements and mandibular movements.

Secondary objectives are the analysis of any correlation between the magnitude of the movement and the airway volume, correlation between the direction of the movements and the changes in airway volume and correlation with Health-Related Quality of Life (HRQoL). Expected confounding factors like smoking habits and Body Mass Index (BMI) will be analyzed.

DETAILED DESCRIPTION:
Background Orthognathic surgery affects the position of the teeth and jaws. The upper airway compartment is in close approximation to these tissues. Consequently, changes of the respiratory volume after surgical treatment in this region is expected.

Orthognathic surgery The correction of severe malocclusions and dentofacial deformities has since the beginning of 20th century been treated with orthodontic and surgical methods. Epidemiologic surveys reveal that about 5 % of the western population has dentofacial disproportions of a magnitude that affect both function and facial aesthetics.

Respiratory disability Obstructive sleep apnea, estimated to occur in between 5% and 10% of the western countries' population. Disabilities in the upper airway may affect the patient's general health and quality of life. Breathing incapability often lead to impaired sleep and consequently decrease the individual's overall capacity and performance. Known predisposing factors are obesity, smoking and age.

Treatment of respiratory disabilities Medical, behavioral and surgical treatment options are prospected methods and the treatment is individually planned in detail. The complex nature of obstructive sleep apnea may require multidisciplinary assessment.

Orthognathic surgery as treatment for obstructive sleep apnea syndrome (OSAS) Correction of anatomical abnormalities may cure obstructive sleep apnea or improve compliance with positive airway pressure treatment. Orthognathic surgery with an anterior movement of the jaws can increase the airway volume and facilitate breathing.

Measurements and evaluation of the upper airway volume Different methods of measuring the upper airway, like physio metric and radiological are present.

Project plan Subjects The study is performed retrospectively on a prospective material. Sixty-two consecutive patients aged between 18 to 30 years with Angle class III occlusion were included in the study.

Patients with systemic diseases in the musculoskeletal apparatus, drug abuse, poor psychic status or disease in the temporomandibular joint were excluded from the study.

Methods The study is performed retrospectively on a prospective material. Examination with clinical examination, BMI, HRQoL questionnaire, dental casts, photography and two- and three-dimensional radiographs and cephalometric measures was performed prior to surgery.

The patient's data (x-ray and photographs) were linked together in computer software programs and used for cephalometric analysis and simulation of the orthodontic and surgical movements (Fasad® and Simplant® PRO 12.00 OMS). The treatment was performed in accordance with this plan.

The last follow up was performed 12 months after surgery including identical registrations as prior to surgery, described above. HRQoL questionnaires consisted of Oral Health Impact Profile (OHIP-S), Jaw Functional Limitation Scale (JFLS-20) and Orofacial Aesthetic Scale (OAS-S). The results from the presurgical questionnaire will be compared with the postsurgical results. Twenty subjects were asked to fill in the follow-up questionnaire twice with two weeks interval for a reliability test of the method.

The pre- and postoperative CT will be compared in a software for measurements of upper airway volume with the software Philips IntelliSpace® Portal, version 11. Measures will be performed with an divided analysis of the upper airway according to the method described by Kim. Thus, the upper airway segmented into four compartments. The measurements will be performed on the sole segment volume and the total airway volume. A comparison of jaw movements, changes in airway volume, BMI and HRQoL will be performed.

Statistical methods The sample size, 62 patients, was based on numbers included in previous similar studies from other centers.

Simple statistics, mean and standard deviation (SD), for all variables will be used. Differences in airway volume and movements, preoperatively and postoperatively will be compared with McNemar's-test. Wilcoxon's paired-sample test will be used for analyzing airway volume before and after surgery as a numeric variable. The reliability test, performed as a test-retest, will be analyzed with the intraclass correlation coefficient, Fisher's test for pair comparisons and Pearson's correlation coefficient. Mann-Whitney-test will be performed to detect differences between questionnaire responses and clinical findings, i.e. BMI, and volumetric findings. The data will be assessed by using Spearman correlation analysis and simple linear regression analysis. Two-sided tests and alpha level 0.05 will be used. Confidence interval (CI) will be calculated. For all computations IBM® SPSS® statistical software will be used.

ELIGIBILITY:
Inclusion Criteria:

* Maxillary retrognatism and Angle class III occlusion deviating at least 5 mm in sagittal and/or vertical aspect from normal occlusion measured as interincisal distance
* Age between 18 to 30 years

Exclusion Criteria:

* Systemic diseases in the musculoskeletal apparatus
* Drug abuse
* Poor psychic status
* Disease in the temporomandibular joint

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Consecutive patients, aged between 18 to 30 years, with diagnosed maxillary retrognatism and Angle class III occlusion deviating at least 5 mm in sagittal and/or vertical aspects from normal occlusion
Sampling Method: Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2021-05-15 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-12-28 (Actual)

PRIMARY OUTCOMES:
Changes in upper airway volume | Preoperative and 12 months postoperative follow up.
  Measurements in three dimensional radiographs from pre- and postoperative recordings.

SECONDARY OUTCOMES:
Correlation BMI and upper airway volume. | Preoperative and 12 months postoperative follow up.
  Correlation between changes in Upper airway volume and Body mass index (BMI).
Direction of surgical movements | Preoperative and 12 months postoperative follow up.
  Correlation between the direction of the surgical movements and the changes of the upper airway volume.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Bengtsson, DDS, PhD, Principal Investigator — Skane University Hospital
Locations (1):
- Dept Oral and Maxillofacial Surgery, Lund, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baldwin CM, Griffith KA, Nieto FJ, O'Connor GT, Walsleben JA, Redline S. The association of sleep-disordered breathing and sleep symptoms with quality of life in the Sleep Heart Health Study. Sleep. 2001 Feb 1;24(1):96-105. doi: 10.1093/sleep/24.1.96. PMID 11204058
- [Background] Moscarino S, Kotter F, Brandt M, Modabber A, Kniha K, Holzle F, Wolf M, Mohlhenrich SC. Influence of different surgical concepts for moderate skeletal class II and III treatment on the nasopharyngeal airway space. J Craniomaxillofac Surg. 2019 Oct;47(10):1489-1497. doi: 10.1016/j.jcms.2019.07.006. Epub 2019 Jul 18. PMID 31399294
- [Background] Kim JS, Kim JK, Hong SC, Cho JH. Pharyngeal airway changes after sagittal split ramus osteotomy of the mandible: a comparison between genders. J Oral Maxillofac Surg. 2010 Aug;68(8):1802-6. doi: 10.1016/j.joms.2009.11.010. Epub 2010 May 26. PMID 20537778
- [Background] Kim YJ, Hong JS, Hwang YI, Park YH. Three-dimensional analysis of pharyngeal airway in preadolescent children with different anteroposterior skeletal patterns. Am J Orthod Dentofacial Orthop. 2010 Mar;137(3):306.e1-11; discussion 306-7. doi: 10.1016/j.ajodo.2009.10.025. PMID 20197163
- [Background] Bengtsson M, Wall G, Greiff L, Rasmusson L. Treatment outcome in orthognathic surgery-A prospective randomized blinded case-controlled comparison of planning accuracy in computer-assisted two- and three-dimensional planning techniques (part II). J Craniomaxillofac Surg. 2017 Sep;45(9):1419-1424. doi: 10.1016/j.jcms.2017.07.001. Epub 2017 Jul 12. PMID 28800842
- [Background] Bengtsson M, Wall G, Miranda-Burgos P, Rasmusson L. Treatment outcome in orthognathic surgery - A prospective comparison of accuracy in computer assisted two and three-dimensional prediction techniques. J Craniomaxillofac Surg. 2018 Nov;46(11):1867-1874. doi: 10.1016/j.jcms.2017.01.035. Epub 2017 Feb 13. PMID 28318923
- [Derived] Pellby D, Bengtsson M. Do Patients Detect Changes in Breathing After Orthognathic Surgery? J Oral Maxillofac Surg. 2024 Jan;82(1):36-46. doi: 10.1016/j.joms.2023.09.017. Epub 2023 Sep 27. PMID 37858599